CLINICAL TRIAL: NCT02638545
Title: Effects of Dexmedetomidine on Pressor Response to Norepinephrine in Patients With Septic Shock
Brief Title: Hemodynamic Effects of Dexmedetomidine in Septic Shock
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Morelli, MD, associate professor, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3820
Record Dates: First submitted 2015-12-18; First posted 2015-12-23 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Sedation with propofol and remifentanyl will be replaced by a sedation with dexmedetomidine and remifentanyl
  Other Names: Dexdor

SUMMARY:
The current treatment regimen of patients with septic shock requires a sufficient hemodynamic support aiming to preserve tissue oxygen requirements and perfusion. Therefore, aggressive fluid challenge and vasopressor agents play a pivotal role. To increase total peripheral resistance and preserve organ perfusion, a continuous infusion of catecholamines is often needed. Because sepsis is usually associated with adrenergic receptor and post-receptor abnormalities, the efficacy of such treatment regimens often gradually decreases over time, thereby complicating hemodynamic support. Experimental evidence suggest that α-2 agonists increase pressor responsiveness following lipopolysaccharide administration. This study will assess the effects of the sedation with dexmedetomidine (α-2 agonist) on norepinephrine requirements in patients with septic shock.

DETAILED DESCRIPTION:
The present study was designed as a prospective study. All patients enrolled in the study will require norepinephrine to maintain MAP between 65 and 75 mmHg despite adequate volume resuscitation and will be sedated according to istitutional guidelines with propofol and remifentanyl. After 8 h had elapsed during stable hemodynamic conditions, an initial set of measurements will be obtained during the sedation with propofol and remifentanyl. This set of measurements will be considered as baseline. In the patients in which conventional sedation will be replaced by dexmedetomidine and remifentanyl, a second set of measurements will be obtained after 4 h had elapsed during stable conditions. A final set of mesurements will be obtained after another 8-h period in stable conditions after switcheing back again to propofol and remifentanyl, .

During the observational period the dosage rate of norepinephrine will be adjusted to maintain the same threshold MAP of 65-75 mmHg All other medications were held constant.

ELIGIBILITY:
Inclusion Criteria:

* septic shock
* need for sedation

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
norepinephrine dose | 4 hours

SECONDARY OUTCOMES:
cardiac output | 4 hours
mean arterial pressure | 4 hours
heart rate | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morelli, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Departement of Anesthesiology and Intensive Care of the University of Rome La Sapienza, Rome, Italy

IPD SHARING:
Plan to Share IPD: No